CLINICAL TRIAL: NCT03317444
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TRC101 in Subjects With Chronic Kidney Disease and Metabolic Acidosis
Brief Title: Evaluation of TRC101 in Subjects With Metabolic Acidosis Associated With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tricida, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRCA-301; 2016-003825-41 (EudraCT Number)
Record Dates: First submitted 2017-10-11; First posted 2017-10-23 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Metabolic Acidosis
Keywords: blood bicarbonate, kidney disease
MeSH Terms: conditions — Acidosis; Kidney Diseases | interventions — veverimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRC101 (Experimental): Administered once daily (QD) for 12 weeks
  Interventions: Drug: TRC101
- Placebo (Placebo Comparator): Administered once daily (QD) for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRC101 — Oral suspension
  Other Names: Veverimer
  Arms: TRC101
Drug: Placebo — Oral suspension
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, placebo-controlled, parallel-design study. The study will enroll approximately 210 adult male and female subjects with stage 3 or 4 chronic kidney disease and metabolic acidosis. The study dosing (TRC101 or placebo) will continue for 12 weeks once daily.

The maximum study duration is anticipated to be up to 16 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Blood bicarbonate level of 12 to 20 mEq/L.
* Estimated glomerular filtration rate (eGFR) of 20 to 40 mL/min/1.73m2.
* Stable kidney function defined as <=20% variability in eGFR during screening period.

Key Exclusion Criteria:

* Any level of low blood bicarbonate during the screening period that in the opinion of the Investigator, requires emergency intervention or evaluation for an acute acidotic process.
* Anuria, dialysis, acute kidney injury, or history of acute kidney insufficiency within 3 months prior to screening.
* Heart failure with maximum New York Heart Association (NYHA) Class IV symptoms or that required hospitalization during the preceding 6 months.
* Heart or kidney transplant.
* Chronic obstructive pulmonary disease (COPD) that is treated with chronic oral steroids, that requires the subject to be on oxygen, or that required hospitalization within the previous 6 months.
* Change in doses to alkali therapy in the 4 weeks prior to screening.
* History or current diagnosis of diabetic gastroparesis, bowel obstruction, swallowing disorders, inflammatory bowel disease, major gastrointestinal surgery, frequent diarrhea or active gastric/duodenal ulcers.
* Serum calcium <= 8.0 mg/dL at screening.
* Planned initiation of renal replacement therapy within 12 weeks following randomization.
* Use of polymeric binder drugs within 14 days prior to screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Tricida, Inc.
Locations (44):
- United States (13):
  - Investigative Site 55, Phoenix, Arizona
  - Investigative Site 56, Chula Vista, California
  - Investigative Site 91, Los Angeles, California
  - Investigative Site 59, Hialeah, Florida
  - Investigative Site 54, Hollywood, Florida
  - Investigative Site 93, Hollywood, Florida
  - Investigative Site 92, Lauderdale Lakes, Florida
  - Investigative Site 51, Tampa, Florida
  - Investigative Site 57, Winter Park, Florida
  - Investigative Site 95, Atlanta, Georgia
  - Investigative Site 53, Shreveport, Louisiana
  - Investigative Site 58, Flushing, New York
  - Investigative Site 52, San Antonio, Texas
- Investigative Site 11, Sofia, Bulgaria
- Investigative Site 21, Zagreb, Croatia
- Georgia (7):
  - Investigative Site 31, Tbilisi
  - Investigative Site 32, Tbilisi
  - Investigative Site 33, Tbilisi
  - Investigative Site 34, Tbilisi
  - Investigative Site 35, Tbilisi
  - Investigative Site 36, Tbilisi
  - Investigative Site 37, Tbilisi
- Hungary (9):
  - Investigative Site 43, Baja
  - Investigative Site 48, Balatonfüred
  - Investigative Site 41, Budapest
  - Investigative Site 46, Budapest
  - Investigative Site 45, Hatvan
  - Investigative Site 49, Hódmezővásárhely
  - Investigative Site 44, Kistarcsa
  - Investigative Site 42, Miskolc
  - Investigative Site 47, Mosonmagyaróvár
- Serbia (4):
  - Investigative Site 64, Belgrade
  - Investigative Site 65, Belgrade
  - Investigative Site 61, Vršac
  - Investigative Site 62, Zrenjanin
- Slovenia (2):
  - Investigative Site 72, Jesenice
  - Investigative Site 71, Maribor
- Ukraine (7):
  - Investigative Site 81, Kharkiv
  - Investigative Site 83, Kharkiv
  - Investigative Site 87, Kharkiv
  - Investigative Site 88, Kharkiv
  - Investigative Site 84, Kyiv
  - Investigative Site 85, Kyiv
  - Investigative Site 86, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wesson DE, Mathur V, Tangri N, Stasiv Y, Parsell D, Li E, Klaerner G, Bushinsky DA. Veverimer versus placebo in patients with metabolic acidosis associated with chronic kidney disease: a multicentre, randomised, double-blind, controlled, phase 3 trial. Lancet. 2019 Apr 6;393(10179):1417-1427. doi: 10.1016/S0140-6736(18)32562-5. Epub 2019 Mar 8. PMID 30857647

RESULTS

PARTICIPANT FLOW:
Groups:
- TRC101 Treatment Arm: The first dose of blinded study drug (2 packets for a total of 6 g TRC101) was given at the study site on Day 1 in the morning with food. For the remainder of the Treatment Period, TRC101 was self-administered orally as an aqueous suspension, QD with lunch, for 12 weeks. Beginning at the Week 4 Visit, subjects could have had a blinded dose adjustment to 0, 3 or 9 g (0, 1 or 3 packets, respectively) of TRC101 QD in accordance with a protocol-specified titration algorithm. The last dose of study drug was to be taken the day before the Week 12 Visit, unless the subject was enrolled in the extension Study TRCA-301E.
- Placebo Treatment Arm: The first dose of blinded study drug (2 packets of placebo) was given at the study site on Day 1 in the morning with food. For the remainder of the Treatment Period, placebo was self-administered orally as an aqueous suspension, QD with lunch, for 12 weeks. Beginning at the Week 4 Visit, subjects could have had a blinded dose adjustment to 0, 1 or 3 packets of placebo QD in accordance with a protocol-specified titration algorithm. The last dose of study drug was to be taken the day before the Week 12 Visit, unless the subject was enrolled in the extension Study TRCA-301E.
Period: Overall Study
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Started | 124 | 93
Completed | 119 | 89
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm | Total
Number analyzed (Participants) | 124 | 93 | 217
Age, Categorical [Count of Participants; unit: Participants] — Age (years) was calculated as the number of years between date of birth and date of informed consent, expressed as an integer.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 59 | 44 | 103
    >=65 years | 65 | 49 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years) was calculated as the number of years between date of birth and date of informed consent, expressed as an integer.
  years | 62.9 (12.64) | 63.3 (12.08) | 63.1 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 33 | 83
  Male | 74 | 60 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 121 | 89 | 210
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
History of Hypertension [Count of Participants; unit: Participants] | 120 | 90 | 210
History of Diabetes Mellitus [Count of Participants; unit: Participants] | 76 | 65 | 141
History of Congestive Heart Failure [Count of Participants; unit: Participants] | 36 | 31 | 67
Baseline Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Baseline eGFR was defined as the average of the values of eGFR collected at the Screening 1 Visit, Screening 2 Visit, and Baseline Visit (i.e., Day 1 pre-dose), based on serum creatinine values measured by the central laboratory and using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
  mL/min/1.73m^2 | 29.2 (6.29) | 27.8 (5.45) | 28.6 (5.97)
Baseline Bicarbonate [Mean (Standard Deviation); unit: mEq/L] — Baseline Bicarbonate was defined as the average of the values of serum bicarbonate collected at the Screening 1 Visit, Screening 2 Visit, and Baseline Visit (i.e., Day 1 pre-dose), measured onsite using an i-STAT point-of-care device.
  mEq/L | 17.27 (1.429) | 17.30 (1.504) | 17.28 (1.458)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Change From Baseline in Serum Bicarbonate of ≥ 4 mEq/L or Serum Bicarbonate Within the Normal Range
Description: Composite endpoint of the percentage of subjects having a change from baseline in serum bicarbonate ≥ 4 mEq/L or having serum bicarbonate in the normal range (22 - 29 mEq/L) at the end of treatment (Week 12 Visit).
Time Frame: Baseline to Week 12
Population: The Modified Intent-to-Treat (MITT) Analysis Set was defined as all randomized subjects who had both baseline and at least one postbaseline serum bicarbonate value measured using an i-STAT device. The MITT Analysis Set was used for evaluation of efficacy, based on planned treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 120 | 89
percentage of participants
  Subjects with change from baseline serum bicarbonate ≥ 4 mEq/L or serum bicarbonate in normal range | 59.2 [49.8 to 68.0] | 22.5 [14.3 to 32.6]
  Subjects with change from baseline serum bicarbonate ≥ 4 mEq/L | 55.8 [46.5 to 64.9] | 21.3 [13.4 to 31.3]
  Subjects with serum bicarbonate in normal range | 50.0 [40.7 to 59.3] | 16.9 [9.8 to 26.3]
Statistical Analysis 1: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; % Subjects Who Met Endpoint (≥ 4 mEq/L Change from Baseline Serum Bicarbonate or Serum Bicarbonate in the Normal Range [22 - 29 mEq/L]): TRC101-Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Treatment difference in % of subjects = 36.7, 95% CI 2-sided [23.5 to 48.9]
Statistical Analysis 2: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; % Subjects with ≥ 4 mEq/L Change from Baseline in Serum Bicarbonate: TRC101-Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Treatment difference in % of subjects = 34.5, 95% CI 2-sided [21.2 to 46.8]
Statistical Analysis 3: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; % Subjects with Serum Bicarbonate in the Normal Range (22 - 29 mEq/L): TRC101-Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Treatment difference in % of subjects = 33.1, 95% CI 2-sided [19.7 to 45.6]

2. Secondary Outcome: Change From Baseline to End of Treatment in Serum Bicarbonate
Description: Mean change from baseline to end of treatment (Week 12 Visit) in serum bicarbonate
Time Frame: Baseline to Week 12
Population: The Modified Intent-to-Treat (MITT) Analysis Set was defined as all randomized subjects who had both baseline and at least one postbaseline serum bicarbonate value measured using an i-STAT device. The MITT Analysis Set was used for evaluation of efficacy, based on planned treatment assignment. For this outcome measure, the analysis was done using a mixed model.
Measure: Least Squares Mean (95% Confidence Interval); unit: mEq/L
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 123 | 93
mEq/L | 4.42 [3.85 to 4.98] | 1.78 [1.13 to 2.44]
Statistical Analysis 1: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; Least Squares (LS) Mean Change from Baseline: TRC101-Placebo; Test type: Superiority; p < 0.0001, Mixed-effect repeated measures model; Treatment difference in LS means = 2.63, 95% CI 2-sided [1.77 to 3.5], Standard Error of Mean 0.44 — Standard error presented above is for the LS mean

ADVERSE EVENTS:
Time Frame: Data are the number of patients with adverse events occurring on or after the date of the first dose of TRC101 or placebo up to 14 weeks.
Groups:
- TRC101 Treatment Arm: The first dose of blinded study drug (2 packets of TRC101 [6 g]) was given at the study site on Day 1 in the morning with food. For the remainder of the Treatment Period, TRC101 was self-administered orally as an aqueous suspension, QD with lunch, for 12 weeks. Beginning at the Week 4 Visit, subjects could have had a blinded dose adjustment to 0, 3 or 9 g (0, 1 or 3 packets, respectively) of TRC101 QD in accordance with a protocol-specified titration algorithm. The last dose of study drug was to be taken the day before the Week 12 Visit, unless the subject was enrolled in the extension Study TRCA-301E.
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/124 | 2/93
Serious Adverse Events (participants affected / at risk) | 3/124 | 2/93
Other Adverse Events (participants affected / at risk) | 31/124 | 13/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC101 Treatment Arm (N=124) | Placebo Treatment Arm (N=93)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC101 Treatment Arm (N=124) | Placebo Treatment Arm (N=93)
Headache (Nervous system disorders) | 7 (7) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 11 (20) | 3 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 (16) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT03317444/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT03317444/SAP_001.pdf